CLINICAL TRIAL: NCT06516822
Title: Circumferential Pulmonary Vein Isolation With Modified Linear Ablation Versus Circumferential Pulmonary Vein Isolation Only in Patients With Long-standing Persistent Atrial Fibrillation (SINUS)
Brief Title: CPVI With Modified Linear Ablation Versus CPVI in Patients With Long-standing Persistent Atrial Fibrillation (SINUS)
Acronym: SINUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhang Fengxiang, Deputy Director of Cardiology, Principal Investigator, Clinical Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-SR-027.A1
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Long-standing Persistent Atrial Fibrillation; Ablation
Keywords: long-standing persistent atrial fibrillation; circumferential pulmonary vein isolation; modified linear ablation; arrhythmia-free survival

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPVI-MLA (Experimental): Patients randomized to the CPVI-MLA group first undergo ethanol infusion in the vein of Marshall (EI-VOM) followed by CPVI, left atrial posterior wall isolation (PWI), linear ablation of mitral isthmus (MI), left atrial intima adjoining CS (LAI-CS) and cavo-tricuspid isthmus (CTI), and superior vena cava isolation (SVCI).
  Interventions: Procedure: CPVI-MLA
- CPVI only (Active Comparator): Patients randomized to the CPVI group undergo right PV ablation, followed by the left PV ablation. Radiofrequency ablation should be applied at least 1-2 cm outside of the PV ostia in a wide-area circumferential pattern. Complete CPVI is achieved when all PV potentials within each antrum recorded by the high-density mapping catheter are abolished.
  Interventions: Procedure: CPVI only

INTERVENTIONS:
Procedure: CPVI-MLA — The details include: (1) EI-VOM procedure: An 8.5-French-long sheath is inserted into to the CS via the femoral vein. A JR4 catheter is inserted into the CS to identify the ostium of the VOM. Subsequently, a guide wire supported by an OTW balloon catheter is advanced into the VOM. The balloon is inflated at 6-8 atm pressure in the VOM. Ethanol is infused into VOM from distal to proximal with 3ml each time within 1-2min. After the distal EI-VOM, the balloon is deflated and adjusted to the middle part of VOM. The EI-VOM procedure in the proximal and middle part of VOM should be the same as that in the distal. After three times of EI-VOM, the contrast is injected into VOM to make it permeable and dispersed to observe the effect of alcohol ablation. (2) After EI-VOM, radiofrequency ablation is performed to achieve bilateral PVI, PWI, bidirectional block of MI and CTI, disappearance of LAI-CS potential and SVCI. (3) Any organized AT observed during the procedure is targeted as well.
  Arms: CPVI-MLA
Procedure: CPVI only — After reconstructing the left atrial geometry, CPVI is performed. Radiofrequency ablation should be applied at least 1-2 cm outside of the PV ostia for PVI to achieve a wide PVI ring. The mapping catheter PentaRay will be used to confirm the complete isolation of the PV antrum when all PV potentials within each antrum are abolished. If the AF persists after CPVI, direct current cardioversion is then be conducted to restore sinus rhythm. If spontaneous AFL/AT occurs during ablation, ablation is performed targeting the focal or critical isthmus under the guidance of high-density activation mapping. The endpoint of CPVI is to achieve complete entrance and exit block of all PV antra as recorded by PentaRay during sinus rhythm or CS pacing.
  Arms: CPVI only

SUMMARY:
Catheter ablation has become as the first-line treatment for patients with symptomatic atrial fibrillation (AF). As the cornerstone of catheter ablation for AF, the safety and efficacy of circumferential pulmonary vein isolation (CPVI) have been confirmed. However, for persistent AF, especially for long-standing persistent AF (LSPAF), the recurrence rate is still high. Whether the ethanol infusion (EI) into the vein of Marshall (EI-VOM) and linear ablation could improve the success rate remains controversial.

The SINUS study is a prospective, multicenter, randomized trial, which is designed to compare the efficacy and safety between CPVI with modified linear ablation (CPVI-MLA) and CPVI only for the treatment of LSPAF.

DETAILED DESCRIPTION:
The SINUS study will include 320 patients with LSPAF undergoing catheter ablation for the first time. All patients will be randomized to either the CPVI-MLA group or CPVI only group in a 1:1 ratio. The CPVI-MLA strategy is a fixed ablation approach consisting of EI-VOM, CPVI, left atrial posterior wall isolation (PWI), linear ablation of mitral isthmus (MI), left atrial intima adjoining CS (LAI-CS) and cavo-tricuspid isthmus (CTI), and superior vena cava isolation (SVCI). The follow-up is for a minimum of 12 months with rhythm monitoring. The primary endpoint is freedom from any documented atrial arrhythmia including atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) > 30 seconds after the initial 3 months blanking period without the use of antiarrhythmic drugs (AADs), at 12 months after the index ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Patients with symptomatic LSPAF refractory to at least one antiarrhythmic drug; LSPAF will be defined as a sustained AF episode lasting ≥ 1 year;
2. AF duration 1-3 years;
3. Age 18 - 75 years;
4. Left atrial diameter (LAD) 43-55 mm on long axis parasternal view;
5. AF recorded within 3 years of enrollment;
6. Patient willing and able to comply with protocol and sign informed consent

Exclusion Criteria:

1. Paroxysmal atrial fibrillation;
2. Persistent AF lasting < 1 year or >3 years;
3. Left atrial thrombosis;
4. Patients with a history of catheter ablation for AF;
5. Patients with severe structural heart disease (severe valvular heart disease, hypertrophic cardiomyopathy, dilated cardiomyopathy, etc.);
6. LAD > 55mm on long axis parasternal view;
7. Left ventricular ejection fraction (LVEF) < 40%;
8. Patients with contraindications to low molecular weight heparin, warfarin or novel oral anticoagulants;
9. One-stop procedure for AF ablation and left atrial appendage occlusion;
10. Alcohol allergy or contrast agent allergy;
11. Patients taking cephalosporin antibiotics within 72 hours prior to ablation;
12. Pulmonary artery systolic pressure > 50mmHg;
13. Patients with unstable angina pectoris;
14. Patients who had undergone percutaneous coronary intervention (PCI) within 3 months;
15. Patients who had undergone surgery within 6 months;
16. Patients ready to receive heart transplantation;
17. Patients with a history of thromboembolism within 6 months;
18. Patients with diagnosed atrial myxoma;
19. Patients with severe respiratory diseases;
20. Patients with infectious diseases in active phase;
21. Patients with poorly controlled systemic immune diseases;
22. Patients with uncured malignant hematological diseases;
23. Patients with uncured malignant solid tumors;
24. Patients with untreated hypothyroidism or hyperthyroidism;
25. Patients with severe liver dysfunction (elevation of transaminases [ALT or AST] >3 times the upper limit of normal range);
26. Patients with end-stage renal failure requiring dialysis;
27. Patients with other serious arrhythmias, such as ventricular tachycardia with hemodynamic instability;
28. Pregnant and lactating women;
29. Patients with psychiatric ailments;
30. BMI < 18.5 or ≥ 30kg/m2;
31. Life expectancy < 2 years;
32. Patients unwilling or unable to give informed consent;
33. Patients unwilling or unable to cooperate to complete follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from any documented atrial arrhythmia off AADs | 12 months
  Freedom from any documented atrial arrhythmia including atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) > 30 seconds assessed by ECG and Holter after the initial 3 months blanking period without the use of antiarrhythmic drugs (AADs), after the index ablation procedure

SECONDARY OUTCOMES:
Freedom from any documented atrial arrhythmia on/off AADs | 12 months
  Freedom from any documented atrial arrhythmia > 30 seconds assessed by ECG and Holter after the initial 3 month blanking period, after the index ablation procedure on/off AADs.
Freedom from any documented AF on/off AADs | 12 months
  Freedom from any documented AF episodes > 30 seconds assessed by ECG and Holter after the initial 3 month blanking period, after the index ablation procedure on/off AADs.
Freedom from any documented AFL/AT on/off AADs | 12 months
  Freedom from any documented AFL/AT episodes > 30 seconds assessed by ECG and Holter after the initial 3 month blanking period, after the index ablation procedure on/off AADs.
AF burden | 12 months
  AF burden (% time) on continuous monitoring during 12 months after the 3-months blanking period.
Freedom from any documented AFL/AT on/off AADs in patients with successful EI-VOM | 12 months
  Freedom from any documented AFL/AT episodes > 30 seconds assessed by ECG and Holter after the initial 3 month blanking period, after the index ablation procedure on/off AADs in patients with successful EI-VOM.
AF burden in patients with successful EI-VOM | 12 months
  AF burden (% time) on continuous monitoring during 12 months after the 3-months blanking period in patients with successful EI-VOM
Freedom from AF/AFL/AT after multiple procedures | 12 months
  Freedom from any documented atrial arrhythmia > 30 seconds assessed by ECG and Holter after the initial 3 month blanking period, after more than one ablation procedure on/off AADs.
Freedom from AF after multiple procedures | 12 months
  Freedom from any documented AF > 30 seconds assessed by ECG and Holter after the initial 3 month blanking period, after more than one ablation procedure on/off AADs.
Freedom from AFL/AT after multiple procedures | 12 months
  Freedom from any documented AFL/AT > 30 seconds assessed by ECG and Holter after the initial 3 month blanking period, after more than one ablation procedure on/off AADs.
AF burden after multiple procedures | 12 months
  AF burden (% time) on continuous monitoring during 12 months (after the 3-months blanking period) after multiple procedures
Hospitalization for cardiovascular disease | 12 months
  Hospitalization for cardiovascular disease (e.g., atrial arrhythmia, heart failure and coronary heart disease)
AFEQT score change between baseline and 12-month | 12 months
  Quality of life assessed by AF effect on quality-of-life (AFEQT) questionnaire
EQ-5D-5L score change between baseline and 12-month | 12 months
  Quality of life assessed by EuroQol 5-dimension (EQ-5D-5L) scale
Incidence of procedural complications | Within 3 months after the procedure
  Cardiac tamponade or perforation, phrenic nerve injury, acute coronary occlusion, death, stroke / thromboembolism related to AF ablation, pulmonary vein stenosis, left atrial oesophageal fistula, and vascular complications requiring intervention (e.g., pseudoaneurysm, arteriovenous fistula).

CONTACTS AND LOCATIONS:
Overall Officials: Fengxiang Zhang, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (10):
- China (10):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University third hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen Hospital, Fuwai Hospital, Chinese Academy of Medical Science, Shenzhen, Guangdong
  - Zhengzhou University People's Hospital, Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - Xijing Hospital, Air Force Medical University, Xi’an, Shanxi
  - Taizhou First People's Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
The data used and analyzed to support the study are available from the principal investigator on reasonable request.